CLINICAL TRIAL: NCT06353360
Title: Tumor-Treating Fields (TTFields) in Combination With Temozolomide and Tislelizumab in The Treatment of Newly Diagnosed Glioblastoma: A Safety and Efficacy Clinical Study
Brief Title: TTField in Combination With Temozolomide and Tislelizumab in The Treatment of Newly Diagnosed Glioblastoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Healthy Life Innovation Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-06
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — tislelizumab; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor Treating Fields + Temozolomide + Tislelizumab (Experimental)
  Interventions: Device: Tumor Treating Fields; Drug: Tislelizumab; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Device: Tumor Treating Fields — Tumor Treating Fields will be administered continuously with a planned ≥ 18 h per day, starting on the Day 1 of cycle 1 (C1D1), throughout the entire course of treatment.
Drug: Tislelizumab — Tislelizumab will be given 300 mg intravenously every 4 weeks beginning on Day 1 of Cycle 2 of adjuvant TMZ. The Tislelizumab treatment should be continued until confirmed PD, unacceptable toxicity, or finished Tislelizumab treatment for other reasons.
Drug: Temozolomide (TMZ) — The patients will carry out 6 cycles of TMZ adjuvant chemotherapy according to the instructions. The dosage of TMZ is 150-200 mg/(m2·d), daily for 5 days followed by 23 days without treatment, the treatment cycle is 28 days. The initial dose of cycle 1 is 150 mg/(m2·d), if patients do not experience TMZ chemotherapy toxicity, the dose should be increased to 200 mg/(m2·d) in subsequent treatment cycles. After 6 cycles of TMZ adjuvant chemotherapy, if the patients do not experience disease progression, it is recommended to continue TMZ adjuvant chemotherapy, or treated according to investigators' recommendations. The TMZ treatment should be continued until confirmed progressive disease (PD), unacceptable toxicity, or finished TMZ treatment for other reasons.

SUMMARY:
The goal of this clinical trial is To investigate the safety and efficacy of Tumor-Treating Fields (TTFields) in combined with temozolomide (TMZ) and tislelizumab in the treatment of newly diagnosed glioblastoma (GBM).

ELIGIBILITY:
Inclusion Criteria:

1. After brain surgery (patients with total resection, partial resection and biopsy were acceptable), the pathological examination confirmed glioblastoma with isocitrate dehydrogenase (IDH) wild-type according to the 2021 World Health Organization (WHO) classification of tumors of the central nervous system.
2. The age of the subjects was ≥18 years old;
3. Supratentorial tumors;
4. Patients who had undergone maximal surgical resection (biopsy) and completed TMZ concurrent chemoradiotherapy were planned for adjuvant TMZ treatment.
5. Karnofsky performance status (KPS) score ≥70;
6. The predicted survival time was ≥3 months.
7. Voluntarily signed informed consent;
8. Subjects of childbearing potential had to agree to use effective contraception for the duration of the trial.

Exclusion Criteria:

1. Early progression of GBM occurred after TMZ+radiation therapy (RT) treatment (except pseudoprogression, imaging examination should be supplemented to further exclude if necessary).
2. The subject had received any other cytotoxic or biologic antineoplastic therapy before enrollment;
3. Distant leptomeningeal metastasis;
4. Patients had a diagnosis of cancer other than glioblastoma and received antineoplastic therapy within 5 years before enrollment, excluding cured stage I prostate cancer, cervical or uterine cancer in situ, breast cancer in situ, and nonmelanoma skin cancer.
5. Previous treatment with anti-PD-1 antibody/anti-PD-L1 antibody and anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody;
6. Participants who had received systemic immunosuppressive therapy (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, or antineoplastic factor agents) within 2 weeks before enrollment. Excluding nasal sprays and inhaled corticosteroids;
7. The presence of an active, known, or suspected autoimmune disease that was judged by the investigator to be unsuitable for this study. The following exclusions may be made: vitiligo, alopecia, Graves' disease, psoriasis, or eczema that did not require systemic treatment within the previous 2 years; Hypothyroidism (due to autoimmune thyroiditis) that is asymptomatic or requires only stable doses of hormone-replacement therapy or type I diabetes that requires only stable doses of insulin-replacement therapy, or childhood asthma that has resolved completely without intervention or recurrence in adulthood without an external trigger.
8. Participants had to meet certain criteria for bone marrow, liver and kidney function before enrollment, and were not eligible if they had any of the following:

   1. Thrombocytopenia (platelet count < 100×103/μL)
   2. Neutropenia (absolute neutrophil count < 1.5×103/μL)
   3. National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) 4 grade non-hematologic toxicity (except alopecia, nausea and vomiting)
   4. Significant liver function impairment -aspartate aminotransferase (AST) or alanine transaminase (ALT) exceeding 3 times the upper limit of normal
   5. Total bilirubin more than 1.5 times the upper limit of the normal range
   6. Severe renal impairment (serum creatinine >1.7 mg/dL, or >150 μmol/L).
9. The subject had an active implanted device (deep brain stimulator, spinal cord stimulator, vagus nerve stimulator, pacemaker, cardiac defibrillator, etc.).
10. Infratentorial tumors;
11. Documented increased intracranial pressure (clinically manifested as severe papilledema, vomiting, nausea, or decreased consciousness);
12. There were infection, ulcer and unhealed wound in the skin where the electrode was applied.
13. A known history of allergy to TMZ or tislelizumab;
14. Skull defects or residual metal fragments in the skull (except titanium plates or nails used for skull surgery);
15. Patients allergic to conductive hydrogels or medical adhesives;
16. Those who are pregnant or preparing to become pregnant or who are breastfeeding;
17. Patients with poor compliance, as judged by the investigator, or other factors considered by the investigator to be not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 18 months
  PFS is defined as the time from the start of treatment until disease progression or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 18 months
  Adverse events will be defined as the incidence, frequency and severity of adverse events (AEs) noted in patients treated with study treatments
Objective response rate (ORR) | Up to 18 months
  ORR is defined as the number (%) of patients with at least 1 visit response of complete response (CR) or partial response (PR).
Disease control rate (DCR) | Up to 18 months
  DCR is defined as the rate of best objective response of CR, PR, or stable disease (SD)
Overall Survival (OS) | Up to 18 months
  OS is defined as the time from the date of treatment until death due to any cause
PFS rate at 6 months | Up to 6 months
  The analysis will be estimated proportions of patients who are progression-free at 6 months following the time of enrollment
PFS rate at 1 year | Up to12 months
  The analysis will be estimated proportions of patients who are progression-free at 1 year following the time of enrollment
OS rate at 1-year | Up to12 months
  The analysis will be estimated proportions of patients who are survival at 1 year following the time of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, China